CLINICAL TRIAL: NCT03552185
Title: Depicting Neurogenic Dysphagia in Multiple Sclerosis Patients; Clinical and Endoscopic Studies
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Shereen M Fathi,MD, professor, Kasr El Aini Hospital
Other Study IDs: SF
Record Dates: First submitted 2018-05-04; First posted 2018-06-11 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
Keywords: Neurogenic Dysphagia; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate neurogenic dysphagia in Multiple Sclerosis patients using dysphagia questionnaires and endoscopic study; and to correlate that to MS types, severity, duration, and imaging modalities

DETAILED DESCRIPTION:
Objectives:

The purpose of this study is to evaluate neurogenic dysphagia in Multiple Sclerosis patients using dysphagia questionnaires and endoscopic study; and to correlate that to MS types, severity, duration, and imaging modalities

Study Design:

Observational, descriptive study

Population of study and disease condition:

Egyptian patients with Clinically Definite Multiple sclerosis according to the MAGNIMS consensus Guidelines and MCdonald's criteria 2017

Selected patients will be all Multiple Sclerosis patients attending Neurology Outpatient Clinic & Neurology Department at Kasr Alainy Hospital within a definite time interval (January 2018- June 2018) with an estimate of 100 patients.

A written consent, approved by the ethical committee of Neurology Department, faculty of medicine, Cairo University will be obtained for each participant.

Methodology in details:

Patients in this study will be submitted to the following:

1. Through history taking and meticulous neurological examination.
2. Clinical & assessment scales:

   1. Expanded Disability status scale (EDSS)
   2. 10-item Dysphagia in Multiple Sclerosis questionnaire (DYMUS): Ten-item questionnaire for assessment of dysphagia in multiple sclerosis. The questionnaire can be divided into two subscales; for the assessment of dysphagia for solids (7 items, in bold), and for the assessment of dysphagia for liquids (3 items, in italics). Instructions for the patient: This questionnaire is about your ability to swallow.
   3. Dysphagia handicap index (DHI): new, easy-to-complete, statistically robust, patient-reported outcomes measure for assessing the handicapping effect of dysphagia. These statements were 60 in number and were sorted into three subscales based on their content. The emotional subscale consisted of 16 statements representing a person's affective response to their dysphagia. There were 27 statements representing a person's self-perception of physical discomfort due to dysphagia. There were 27 statements representing a person's self-perception of physical discomfort due to dysphagia. In order to evaluate an overall picture of the patient's perception of their dysphagia, all subscales were combined to provide an overall total DHI score. At the completion of the test, subjects were asked to self-rate the severity of their dysphagia on a 7-point equal appearing interval scale.
3. Flexible Endoscopic Evaluation of Swallowing (FEES): will be performed to MS patients with dysphagia as detected by dysphagia questionnaires.
4. Neuro-imaging: Magnetic Resonance imaging of the brain and spinal cord with contrast were performed for patients on a 1.5 Tesla Phillips Intera® Scanner at the Magnetic Resonance unit, Department of Radio-diagnosis, Cairo University. The following protocols were used:

   * T1-weighted images (axial & sagittal)
   * T2-weighted images (axial & coronal)
   * Fluid attenuated inversion recovery (FLAIR) sequence

Correlation of endoscopy result with type of MS (whether RRMS or progressive form), severity of disease (as assessed by EDSS), duration of disease (number of years since first symptom), and lesion load (assessed by MRI)

Possible Risk:

Uncommon complications of FEES as epistaxis and vasovagal attack (very rare).

Primary outcomes:

To screen the prevalence of neurogenic dysphagia in Egyptian MS patients attending Neurology Outpatient Clinic & Neurology Department at Kasr Alainy Hospital within a definite time interval( January 2018 - June 2018)

Secondary outcome parameters (other outcomes to be assessed) To depict neurogenic dysphagia in MS and assessment of its efficiency as a biomarker for disease progression.

Statistical analysis:

Results will be evaluated statistically by Statistical Package for the Social Sciences "SPSS" version 16.

Data will be summarized using mean and standard deviation for quantitative variables and percent for qualitative variables.

Comparison between groups will be done using chi square test for quantitative variables & ANOVA (analysis of variance).

Multiple comparisons will be done using post Hoc test for normally distributed quantitative variables and parametrical. Mann-Whitney test for not normally distributed quantitative variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Multiple Sclerosis

Exclusion Criteria:

* Local causes of Dysphagia excluded by proper history taking, proper clinical examination (e.g.; esophageal tumor, GERD, Achalasia, Radiation therapy)
* Anatomical changes in the oral cavity, pharynx and larynx that might interfere with swallowing (i.e.: , history of recent trauma to the nasal cavity or surrounding tissue )
* Patients with tracheostomy or a history of having been submitted to it.
* Patients with contraindications of Flexible Endoscopic Evaluation of Swallowing as severe dyskinesia.
* Severe bleeding disorders and/or recent severe epistaxis, and bilateral obstruction of the nasal passages.
* History of major systemic disease e.g.; renal, hepatic, thyroid diseases, and collagen vascular disorders.
* Non cooperative patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Egyptian patients with Clinically Definite Multiple sclerosis according McDonald's criteria 2017
  Selected patients will be all Multiple Sclerosis patients attending Neurology Outpatient Clinic & Neurology Department at Kasr Alainy Hospital within a definite time interval (January 2018- June 2018) with an estimate of 100 patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
screen the prevalence of neurogenic dysphagia in Egyptian MS patients attending Kasr Alainy hospital during specified peroid of time using validated dysphagia Questionnaires | January 2018 - June 2018
  To screen the prevalence of neurogenic dysphagia in Egyptian MS patients attending Neurology Outpatient Clinic & Neurology Department at Kasr Alainy Hospital within a definite time interval using Ten-item questionnaire for assessment of dysphagia in multiple sclerosis (DYMUS). The higher the score the more or worse dysphagia. the score range from 0 - 10. Patient scored 3 or more on DYMUS questionnaire considered to have dysphagia
screen the prevalence of neurogenic dysphagia in Egyptian MS patients attending Kasr Alainy hospital during specified peroid of time using validated dysphagia Questionnaires | January 2018 - June 2018
  To screen the prevalence of neurogenic dysphagia in Egyptian MS patients having dysphagia by questionnaires attending Neurology Outpatient Clinic & Neurology Department at Kasr Alainy Hospital within a definite time interval using Dysphagia handicap index (DHI). The higher the score the more or worse dysphagia. the score range from 1 - 7. no cut off value
Assessment of neurogenic dysphagia in Egyptian MS patients attending Kasr Alainy hospital during specified peroid of time using validated dysphagia Questionnaires | January 2018 - June 2018
  To assess severity/degree of neurogenic dysphagia in Egyptian MS patients attending Neurology Outpatient Clinic & Neurology Department at Kasr Alainy Hospital within a definite time interval using Flexible Endoscopic Evaluation of Swallowing (FEES) for MS patients with dysphagia. it measures degree of dysphagia endoscopically, and the higher the score the more or worse dysphagia. no cut off value. the score range from 1 - 15.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided